

Mann-Whitney tests were conducted for the quantitative and qualitative assessments to identify any significant differences between the 2 doses of ICG. A 2-way ANOVA was also conducted to compare the individual fluorescence intensities of the liver, bile duct, and background fat between the 2 doses. A p value of <0.05 was considered statistically significant. All tests were performed using GraphPad Prism software version 9.4.1 (GraphPad Software, San Diego, CA). Power analysis based on results from our previous study indicated that a total of 26 patients (13 in each arm) would be required for 90% power to detect a difference in the primary outcome measure of bile duct—to—liver fluorescence intensity ratio of 0.2 between the 2 groups, given an alpha of 0.05 and a SD of 0.15. We therefore powered the study to allow for accrual of adequate numbers of subjects at each center independently.